CLINICAL TRIAL: NCT04138329
Title: Comparison of Postoperative Inguinal Pain Between the Onstep Technique and the Lichtenstein Technique: A Randomized Controlled Study.
Brief Title: Comparison of Postoperative Inguinal Pain Between the Onstep Technique and the Lichtenstein Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Principal Investigator, JORGE AGUILAR GARCIA, Surgeon at the General Surgery Department, Hospital Central "Dr. Ignacio Morones Prieto"
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 48-18
Record Dates: First submitted 2019-10-21; First posted 2019-10-24 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Chronic Pain Post-Procedural

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lichtenstein Technique (Active Comparator): In this arm the inguinal hernia repair was made with the Lichtenstein technique by surgeons with experience in this kind of plasty using the conventional polypropylene mesh.
  Interventions: Procedure: Lichtenstein Technique
- Onstep Technique (Experimental): In this arm the inguinal hernia repair was made with the Onstep technique by one surgeon with experience using the Bard's 3DMAX mesh.
  Interventions: Procedure: Onstep Technique

INTERVENTIONS:
Procedure: Lichtenstein Technique — In this group was used the Lichtenstein technique for inguinal repair
  Arms: Lichtenstein Technique
Procedure: Onstep Technique — In this group was used the Onstep technique for inguinal repair
  Arms: Onstep Technique

SUMMARY:
This is a randomized, double blind, controlled study. The aim is to compare postoperative inguinal pain using the Inguinal Pain Questionnaire (IPQ) validated in Spanish and Numerical Pain Scale in postoperative patients with Lichtenstein and Onstep technique at 1 week, 1, 3 and 6 months. The investigators also validated the IPQ in spanish. It was randomized 20 patients for the Lichtenstein repair and 20 patients for the Onstep technique. The study was conducted in the General Surgery Department of the Central Hospital Dr. Ignacio Morones Prieto, considered as a second level of attention and a surgery training center. The validated questionnaire in spanish and the visual pain scale were applied in the office at 1 week and by phone at 1 month, 3 and 6 months after surgery by two evaluators who did not know the surgical technique used.

DETAILED DESCRIPTION:
The investigators use the Browne method to estimate the number of patients required for the study. It was applied simple randomization of 40 patients in two groups, the first one consists of 20 patients for the Lichtenstein repair and the second group of 20 patients for Onstep repair.

The Onstep procedure was performed by a surgeon skilled in the technique as described in the original article by Rosenberg and 3DMAXTM mesh by Bard was used. The technique is simple, the duration of the surgery is short and consists of a series of standardized steps. It combines an anterior with a preperitoneal approach, consisting of making a lateral incision to the rectus abdominis muscle and above the inguinal canal. It is dissected to a plane between the external and internal oblique fascia, the spermatic cord is dissected and sac reduction is performed, either directly or indirectly. The transversalis fascia is incised and the preperitoneal space is dissected. The mesh is preformed laterally to reinforce the deep inguinal ring and medially accommodates in the previously dissected preperitoneal space. The mesh was fixed to the Cooper's ligament, the pubic tubercle and the rectus abdominis muscle with 2-0 polypropylene suture.

The Lichtenstein technique was performed by different surgeons and regular polypropylene mesh was used.

The validated questionnaire in spanish and the visual pain scale were applied in the office at 1 week and by phone at 1 month, 3 and 6 months after surgery by two evaluators who did not know the surgical technique used. Statistical analysis of the results of the survey and visual pain scale in patients operated with the Onstep and Lichtenstein technique was performed with Student's t test and Fisher's exact test.

For the validation of the Inguinal Pain Questionnaire in our population the English-Spanish translation of the IPQ was carried out. Then the translation from Spanish to English was made by a person with English proficiency adjusting the initial translation. All postoperative patients with unilateral inguinal plasty, older than 16 years, with Lichtenstein or laparoscopic technique (TEP and TAPP), performed by different surgeons were included. The survey was applied in Spanish and numerical scale of pain to 21 patients who met the inclusion criteria, operated at the Central Hospital "Dr. Ignacio Morones Prieto", a week and a month after surgery. The first survey was conducted in the first week after surgery, the second was applied by telephone 4 weeks later, both performed by evaluators familiarized with the survey and unrelated to the knowledge of the surgical technique used. Analysis of the survey data was carried out using Cronbach's alpha for internal validation, re-test with the Spearman's rho to compare the variability of the responses with time and finally, the answers of the survey were compared with the score of the numerical scale of pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unilateral inguinal hernia.
* Male or Female.
* Older tan 16 years.
* Accept to participate in the study.

Exclusion Criteria:

* Chronic Obstructive Pulmonary Disease.
* Obesity.
* Diabetes Mellitus.
* Cirrhosis.
* Diseases involving collagen deficiency.
* Previous surgery in the groin.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-03-24 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Postoperative inguinal pain assessed by the Inguinal Pain Questionnaire validated in spanish. | The questionnaire was applied at 1 week after surgery
  The inguinal pain questionnaire (IPQ) was developed by U. Fränneby et al. and published in 2008 as a tool to measure pain behavior. Evaluates the current inguinal pain, the worst pain experienced in the last week and interference with daily activities due to pain. There is a total of 18 questions with a duration of less than 10 minutes to complete it. They concluded that the questionnaire produces valid and reliable information on the frequency and severity of inguinal pain. The investigators also validated this survey in spanish so it could be applied in the study population.
Postoperative inguinal pain assessed by the Inguinal Pain Questionnaire validated in spanish. | The questionnaire was applied at 1 month after surgery
  The inguinal pain questionnaire (IPQ) was developed by U. Fränneby et al. and published in 2008 as a tool to measure pain behavior. Evaluates the current inguinal pain, the worst pain experienced in the last week and interference with daily activities due to pain. There is a total of 18 questions with a duration of less than 10 minutes to complete it. They concluded that the questionnaire produces valid and reliable information on the frequency and severity of inguinal pain. The investigators also validated this survey in spanish so it could be applied in the study population.
Postoperative inguinal pain assessed by the Inguinal Pain Questionnaire validated in spanish. | The questionnaire was applied at 3 months after surgery
  The inguinal pain questionnaire (IPQ) was developed by U. Fränneby et al. and published in 2008 as a tool to measure pain behavior. Evaluates the current inguinal pain, the worst pain experienced in the last week and interference with daily activities due to pain. There is a total of 18 questions with a duration of less than 10 minutes to complete it. They concluded that the questionnaire produces valid and reliable information on the frequency and severity of inguinal pain. The investigators also validated this survey in spanish so it could be applied in the study population.
Postoperative inguinal pain assessed by the Inguinal Pain Questionnaire validated in spanish. | The questionnaire was applied at 6 months after surgery
  The inguinal pain questionnaire (IPQ) was developed by U. Fränneby et al. and published in 2008 as a tool to measure pain behavior. Evaluates the current inguinal pain, the worst pain experienced in the last week and interference with daily activities due to pain. There is a total of 18 questions with a duration of less than 10 minutes to complete it. They concluded that the questionnaire produces valid and reliable information on the frequency and severity of inguinal pain. The investigators also validated this survey in spanish so it could be applied in the study population.
Postoperative inguinal pain assessed by Numerical Pain Rating Scale | The scale was applied at 1 week after surgery
  This scale is a segmented numeric version of the visual analog scale in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of pain, 0 means no pain and 10 the worst pain ever.
Postoperative inguinal pain assessed by Numerical Pain Rating Scale | The scale was applied at 1 month after surgery
  This scale is a segmented numeric version of the visual analog scale in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of pain, 0 means no pain and 10 the worst pain ever.
Postoperative inguinal pain assessed by Numerical Pain Rating Scale | The scale was applied at 3 months after surgery
  This scale is a segmented numeric version of the visual analog scale in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of pain, 0 means no pain and 10 the worst pain ever.
Postoperative inguinal pain assessed by Numerical Pain Rating Scale | The scale was applied at 6 months after surgery
  This scale is a segmented numeric version of the visual analog scale in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of pain, 0 means no pain and 10 the worst pain ever.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Aguilar García, Principal Investigator — Hospital Central "Dr. Ignacio Morones Prieto"
Locations (1):
- Hospital Central Dr. Ignacio Morones Prieto, San Luis Potosí City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenberg J, Andresen K. The Onstep Method for Inguinal Hernia Repair: Operative Technique and Technical Tips. Surg Res Pract. 2016;2016:6935167. doi: 10.1155/2016/6935167. Epub 2016 Jun 9. PMID 27379255
- [Background] Andresen K, Burcharth J, Fonnes S, Hupfeld L, Rothman JP, Deigaard S, Winther D, Errebo MB, Therkildsen R, Hauge D, Sorensen FS, Bjerg J, Rosenberg J. Chronic pain after inguinal hernia repair with the ONSTEP versus the Lichtenstein technique, results of a double-blinded multicenter randomized clinical trial. Langenbecks Arch Surg. 2017 Mar;402(2):213-218. doi: 10.1007/s00423-016-1532-y. Epub 2016 Nov 11. PMID 27837273
- [Background] Alfieri S, Amid PK, Campanelli G, Izard G, Kehlet H, Wijsmuller AR, Di Miceli D, Doglietto GB. International guidelines for prevention and management of post-operative chronic pain following inguinal hernia surgery. Hernia. 2011 Jun;15(3):239-49. doi: 10.1007/s10029-011-0798-9. Epub 2011 Mar 2. PMID 21365287
- [Background] Franneby U, Gunnarsson U, Andersson M, Heuman R, Nordin P, Nyren O, Sandblom G. Validation of an Inguinal Pain Questionnaire for assessment of chronic pain after groin hernia repair. Br J Surg. 2008 Apr;95(4):488-93. doi: 10.1002/bjs.6014. PMID 18161900
- [Background] Lourenco A, da Costa RS. The ONSTEP inguinal hernia repair technique: initial clinical experience of 693 patients, in two institutions. Hernia. 2013 Jun;17(3):357-64. doi: 10.1007/s10029-013-1057-z. Epub 2013 Feb 24. PMID 23435639
- [Background] Aasvang E, Kehlet H. Chronic postoperative pain: the case of inguinal herniorrhaphy. Br J Anaesth. 2005 Jul;95(1):69-76. doi: 10.1093/bja/aei019. Epub 2004 Nov 5. No abstract available. PMID 15531621
- [Background] Browne RH. On the use of a pilot sample for sample size determination. Stat Med. 1995 Sep 15;14(17):1933-40. doi: 10.1002/sim.4780141709. PMID 8532986
- [Derived] Aguilar-Garcia J, Villafuerte-Fernandez R, Ntezes-Hidalgo PI, Meade-Aguilar JA, Ramirez-GarciaLuna JL, Martinez-Jimenez MA. Postoperative inguinal pain and disability after Lichtenstein versus ONSTEP hernia repair: analysis of responses to the inguinal pain questionnaire in Spanish. Surg Today. 2021 May;51(5):703-712. doi: 10.1007/s00595-020-02155-8. Epub 2020 Oct 11. PMID 33040236